CLINICAL TRIAL: NCT01618916
Title: A Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3015014 in Japanese and Non-Japanese Subjects With Elevated LDL-C
Brief Title: A Study of LY3015014 in Otherwise Healthy Participants With High Low-density Lipoprotein (LDL) Cholesterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14354; I5S-EW-EFJB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — frovocimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1.0 milligrams per kilogram (mg/kg) LY3015014 Every 2 Weeks (Experimental): 1.0 mg/kg LY3015014 given subcutaneously (SC) once every 2 weeks for 29 days.
  Interventions: Drug: LY3015014
- 1.0 mg/kg LY3015014 Every 4 Weeks (Experimental): 1.0 mg/kg LY3015014 given SC once every 4 weeks for 29 days.
  Interventions: Drug: LY3015014
- 3.0 mg/kg LY3015014 Every 2 Weeks (Experimental): 3.0 mg/kg LY3015014 given SC once every 2 weeks for 29 days.
  Interventions: Drug: LY3015014
- 3.0 mg/kg LY3015014 Every 4 Weeks (Experimental): 3.0 mg/kg LY3015014 given SC once every 4 weeks for 29 days.
  Interventions: Drug: LY3015014
- Placebo Every 2 Weeks (Placebo Comparator): Saline injection (to match LY3015014) given SC once every 2 weeks for 29 days.
  Interventions: Other: Placebo
- Placebo Every 4 Weeks (Placebo Comparator): Saline injection (to match LY3015014) given SC once every 4 weeks for 29 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LY3015014 — Administered SC
  Arms: 1.0 mg/kg LY3015014 Every 4 Weeks; 1.0 milligrams per kilogram (mg/kg) LY3015014 Every 2 Weeks; 3.0 mg/kg LY3015014 Every 2 Weeks; 3.0 mg/kg LY3015014 Every 4 Weeks
Other: Placebo — Administered SC
  Arms: Placebo Every 2 Weeks; Placebo Every 4 Weeks

SUMMARY:
This is a phase 1 study in otherwise healthy participants with high LDL cholesterol. Following multiple doses of LY3015014, the safety and tolerability of the drug, how the body handles the drug, and the drug's effect on the body will be evaluated. Participants will participate in the study for approximately 3 months not including screening. Screening is required within 42 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy males or females without childbearing potential as determined by medical history and physical examination, including first-generation Japanese participants
* Have body mass indexes of 18 to 35 kilograms per meter square (kg/m^2), inclusive, at screening
* Have screening low-density lipoprotein cholesterol (LDL-C) of between 100 and 180 milligrams per deciliter (mg/dL), inclusive

Exclusion Criteria:

* Have known allergies to compounds related to LY3015014 or any components of the formulation or known clinically significant hypersensitivity to biologic agents
* Have a history of atopy, significant allergies to humanized monoclonal antibodies, clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe posttreatment hypersensitivity reactions [including but not limited to erythema multiforme major, linear immunoglobulin (Ig)A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis)
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, of constituting a risk when taking the study medication, or of interfering with the interpretation of data
* Have received any vaccine(s) within 1 month of LY3015014 dosing or intend to do so during the study
* Have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 1.0 mg/kg LY3015014 Q2W: LY3015014: 1.0 milligrams per kilogram (mg/kg) given as subcutaneous (SC) injection every 2 weeks (Q2W) on Days 1, 15, and 29 for a total of 3 doses.
- 1.0 mg/kg LY3015014 Q4W: LY3015014: 1.0 mg/kg given as SC injection every 4 weeks (Q4W) on Days 1 and 29 for a total of 2 doses.
- 3.0 mg/kg LY3015014 Q2W: LY3015014: 3.0 mg/kg given as SC injection Q2W on Days 1, 15, and 29 for a total of 3 doses.
- 3.0 mg/kg LY3015014 Q4W: LY3015014: 3.0 mg/kg given as SC injection Q4W on Days 1 and 29 for a total of 2 doses.
- Placebo Q2W: Placebo given as SC injection Q2W on Days 1, 15, and 29 for a total of 3 doses.
- Placebo Q4W: Placebo given as SC injection Q4W on Days 1 and 29 for a total of 2 doses.
Period: Overall Study
Arm/Group | 1.0 mg/kg LY3015014 Q2W | 1.0 mg/kg LY3015014 Q4W | 3.0 mg/kg LY3015014 Q2W | 3.0 mg/kg LY3015014 Q4W | Placebo Q2W | Placebo Q4W
Started | 12 | 10 | 11 | 9 | 5 | 4
Received At Least 1 Dose of Study Drug | 12 | 10 | 11 | 9 | 5 | 4
Completed | 10 | 9 | 10 | 7 | 4 | 4
Not Completed | 2 | 1 | 1 | 2 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug (LY3015014 or placebo).
Groups:
- 1.0 mg/kg LY3015014 Q2W: LY3015014: 1.0 mg/kg given as SC injection Q2W on Days 1, 15, and 29 for a total of 3 doses.
- 1.0 mg/kg LY3015014 Q4W: LY3015014: 1.0 mg/kg given as SC injection Q4W on Days 1 and 29 for a total of 2 doses.
- Total: Total of all reporting groups
Arm/Group | 1.0 mg/kg LY3015014 Q2W | 1.0 mg/kg LY3015014 Q4W | 3.0 mg/kg LY3015014 Q2W | 3.0 mg/kg LY3015014 Q4W | Placebo Q2W | Placebo Q4W | Total
Number analyzed (Participants) | 12 | 10 | 11 | 9 | 5 | 4 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (8.0) | 46.8 (10.3) | 53.7 (11.6) | 51.4 (13.6) | 49.2 (13.2) | 47.8 (15.2) | 50.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9 | 3 | 2 | 2 | 25
  Male | 6 | 7 | 2 | 6 | 3 | 2 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 4 | 3 | 3 | 1 | 0 | 16
  Black or African American | 4 | 3 | 3 | 2 | 3 | 2 | 17
  White | 3 | 3 | 5 | 4 | 1 | 1 | 17
  Multiple | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 10 | 11 | 9 | 5 | 4 | 51
Baseline Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 139.6 (26.1) | 119.3 (48.1) | 141.8 (20.2) | 151.7 (30.6) | 165.0 (28.9) | 122.7 (36.0) | 139.4 (33.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Drug Related Treatment-Emergent Adverse Events (TEAEs) or Any Serious AEs (SAEs)
Description: TEAEs were defined as SAEs and other non-serious AEs that occurred or worsened after study treatment. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events section of this report.
Time Frame: Baseline through study completion (up to Day 127)
Population: All enrolled participants who received at least 1 dose of study drug (LY3015014 or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Q2W Plus Placebo Q4W: Placebo given as SC injection Q2W on Days 1, 15, and 29 for a total of 3 doses and Q4W on Days 1 and 29 for a total of 2 doses.
Arm/Group | 1.0 mg/kg LY3015014 Q2W | 1.0 mg/kg LY3015014 Q4W | 3.0 mg/kg LY3015014 Q2W | 3.0 mg/kg LY3015014 Q4W | Placebo Q2W Plus Placebo Q4W
Number analyzed (Participants) | 12 | 10 | 11 | 9 | 9
Participants
  1 or More TEAEs Related to Study Drug | 4 | 3 | 5 | 2 | 3
  Any SAEs | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3015014
Description: The Cmax following the first dose and last dose of LY3015014 is reported.
Time Frame: First Dose (Day 1) and Last Dose (Day 29): Predose, 4 Hours and 24 Hours Postdose
Population: All randomized participants who received at least 1 dose of LY3015014 and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | 1.0 mg/kg LY3015014 Q2W | 1.0 mg/kg LY3015014 Q4W | 3.0 mg/kg LY3015014 Q2W | 3.0 mg/kg LY3015014 Q4W
Number analyzed (Participants) | 12 | 10 | 10 | 9
micrograms per milliliter (µg/mL)
  First Dose | 4.24 (59) | 4.82 (53) | 14.6 (48) | 17.9 (61)
  Last Dose: number analyzed (Participants) | 11 | 10 | 10 | 9
  Last Dose | 9.21 (38) | 6.64 (31) | 35.1 (24) | 23.1 (51)

3. Secondary Outcome: PK: Area Under the Concentration Curve of LY3015014 During 1 Dosing Interval (AUC[0-tau])
Description: The AUC(0-tau) following the first dose and last dose of LY3015014 is reported.
Time Frame: First Dose (Day 1) and Last Dose (Day 29): Predose, 4 Hours and 24 Hours Postdose
Population: All randomized participants who received at least 1 dose of LY3015014 and had evaluable AUC(0-tau) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter (µg*h/mL)
Arm/Group | 1.0 mg/kg LY3015014 Q2W | 1.0 mg/kg LY3015014 Q4W | 3.0 mg/kg LY3015014 Q2W | 3.0 mg/kg LY3015014 Q4W
Number analyzed (Participants) | 12 | 10 | 10 | 9
micrograms*hours/milliliter (µg*h/mL)
  First Dose | 1080 (51) | 2110 (37) | 3890 (47) | 8230 (52)
  Last Dose: number analyzed (Participants) | 11 | 10 | 10 | 9
  Last Dose | 2450 (35) | 2810 (24) | 9440 (17) | 10900 (44)

4. Secondary Outcome: PK: Time of Maximum Concentration (Tmax) of LY3015014
Description: The tmax following the first dose and last dose of LY3015014 is reported.
Time Frame: First Dose: Predose (Day 1) up to Week 4 postdose and Last Dose: predose (Day 29) up to Week 14 postdose
Population: All randomized participants who received at least 1 dose of LY3015014 and had evaluable tmax data.
Measure: Median (Full Range); unit: days
Arm/Group | 1.0 mg/kg LY3015014 Q2W | 1.0 mg/kg LY3015014 Q4W | 3.0 mg/kg LY3015014 Q2W | 3.0 mg/kg LY3015014 Q4W
Number analyzed (Participants) | 12 | 10 | 10 | 9
days
  First Dose | 4 [4 to 14] | 4 [4 to 14] | 4 [1 to 14] | 4 [4 to 14]
  Last Dose: number analyzed (Participants) | 11 | 10 | 10 | 9
  Last Dose | 5 [0 to 5] | 5 [5 to 6] | 5 [5 to 5] | 5 [5 to 14]

5. Secondary Outcome: Percent Change From Baseline to Days 43, 57, and 127 in LDL-C
Description: Percent change from baseline in LDL-C was calculated as Least Squares (LS) mean using mixed effect model repeated measures (MMRM) analysis adjusted for baseline measurement, treatment, day after dosing, and treatment by day interaction.
Time Frame: Baseline, Day 43, Day 57, and Day 127
Population: Randomized participants who received at least 1 dose of study drug (LY3015014 or placebo) and had a baseline and at least 1 postbaseline measurement for LDL-C.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | 1.0 mg/kg LY3015014 Q2W | 1.0 mg/kg LY3015014 Q4W | 3.0 mg/kg LY3015014 Q2W | 3.0 mg/kg LY3015014 Q4W | Placebo Q2W Plus Placebo Q4W
Number analyzed (Participants) | 10 | 9 | 10 | 7 | 9
percentage of change
  Day 43 | -49.76 [-56.71 to -42.81] | -47.56 [-55.30 to -39.82] | -45.20 [-53.69 to -36.70] | -46.64 [-54.66 to -38.62] | 0.16 [-11.88 to 12.20]
  Day 57 | -47.01 [-53.96 to -40.06] | -44.41 [-52.25 to -36.57] | -44.20 [-52.69 to -35.70] | -56.80 [-64.81 to -48.78] | -12.16 [-24.20 to -0.12]
  Day 127 | -7.52 [-14.57 to 0.47] | -15.09 [-22.93 to -7.25] | -23.39 [-31.89 to -14.90] | -18.91 [-27.24 to -10.59] | -0.99 [-13.03 to 11.05]
Statistical Analysis 1: Comparison: 1.0 mg/kg LY3015014 Q2W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis; P-value is for Day 43; Mean Difference (Net) = -49.92, 90% CI [-63.84 to -35.99]
Statistical Analysis 2: Comparison: 1.0 mg/kg LY3015014 Q2W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis; P-value is for Day 57; Mean Difference (Net) = -34.85, 90% CI [-48.78 to -20.93]
Statistical Analysis 3: Comparison: 1.0 mg/kg LY3015014 Q4W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis; P-value is for Day 43; Mean Difference (Net) = -47.72, 90% CI [-62.10 to -33.34]
Statistical Analysis 4: Comparison: 1.0 mg/kg LY3015014 Q4W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis; P-value is for Day 57; Mean Difference (Net) = -32.26, 90% CI [-46.69 to -17.82]
Statistical Analysis 5: Comparison: 3.0 mg/kg LY3015014 Q2W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis; P-value is for Day 43; Mean Difference (Net) = -45.36, 90% CI [-60.07 to -30.64]
Statistical Analysis 6: Comparison: 3.0 mg/kg LY3015014 Q2W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis; P-value is for Day 57; Mean Difference (Net) = -32.04, 90% CI [-46.76 to -17.32]
Statistical Analysis 7: Comparison: 3.0 mg/kg LY3015014 Q4W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis; P-value is for Day 43; Mean Difference (Net) = -46.80, 90% CI [-61.12 to -32.49]
Statistical Analysis 8: Comparison: 3.0 mg/kg LY3015014 Q4W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Analysis; P-value is for Day 57; Mean Difference (Net) = -44.64, 90% CI [-58.95 to -30.32]
Statistical Analysis 9: Comparison: 1.0 mg/kg LY3015014 Q2W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p = 0.440, Mixed Effect Model Analysis; P-value is for Day 127; Mean Difference (Net) = -6.53, 90% CI [-20.51 to 7.44]
Statistical Analysis 10: Comparison: 1.0 mg/kg LY3015014 Q4W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p = 0.108, Mixed Effect Model Analysis; P-value is for Day 127; Mean Difference (Net) = -14.10, 90% CI [-28.53 to 0.33]
Statistical Analysis 11: Comparison: 3.0 mg/kg LY3015014 Q2W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p = 0.013, Mixed Effect Model Analysis; P-value is for Day 127; Mean Difference (Net) = -22.41, 90% CI [-37.13 to -7.69]
Statistical Analysis 12: Comparison: 3.0 mg/kg LY3015014 Q4W vs Placebo Q2W Plus Placebo Q4W; Test type: Superiority or Other; p = 0.042, Mixed Effect Model Analysis; P-value is for Day 127; Mean Difference (Net) = -17.93, 90% CI [-32.42 to -3.44]

ADVERSE EVENTS:
Arm/Group | 1.0 mg/kg LY3015014 Q2W | 1.0 mg/kg LY3015014 Q4W | 3.0 mg/kg LY3015014 Q2W | 3.0 mg/kg LY3015014 Q4W | Placebo Q2W | Placebo Q4W
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/11 | 0/9 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 7/12 | 6/10 | 8/11 | 7/9 | 3/5 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.0 mg/kg LY3015014 Q2W (N=12) | 1.0 mg/kg LY3015014 Q4W (N=10) | 3.0 mg/kg LY3015014 Q2W (N=11) | 3.0 mg/kg LY3015014 Q4W (N=9) | Placebo Q2W (N=5) | Placebo Q4W (N=4)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/6 (0) | 0/3 (0) | 1/9 (1) | 0/3 (0) | 0/2 (0) | 0/2 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0/6 (0) | 1/3 (1) | 0/9 (0) | 0/3 (0) | 0/2 (0) | 0/2 (0)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days